CLINICAL TRIAL: NCT01525381
Title: Strategies to Improve Diagnosis and Treatment of Asthma in Canadians
Brief Title: Strategies to Improve Asthma and Treatment of Asthma in Canadians
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-221
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our study will enroll 644 randomly-selected Canadians who have been diagnosed with asthma by a physician within the previous five years. It will be determined what diagnostic tests were initially performed to make this diagnosis. Participants will undergo lung function testing over 6-8 weeks to determine their respiratory status and to confirm they have asthma. Participants may be followed up to one year depending on their test results.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a recent diagnosis of asthma by a physician. Diagnosis of asthma must have occurred within 5 years prior to entry into the study.
2. Patient must be at least 18 years old.

Exclusion Criteria:

1. Patients in whom methacholine challenge is contraindicated

   * Patients using chronic oral prednisone.
   * Patients with heart attack or stroke within three previous months, and those with known aortic or cerebral aneurysms.
   * Pregnant patients (unknown effect of methacholine on the fetus) and breastfeeding patients (unknown whether methacholine is excreted in breast milk).
2. Patients unable to provide informed consent.
3. Patients not able to perform spirometry and/or methacholine challenge testing.
4. Patients who have a greater than 10 pack-year smoking history (this will exclude patients with possible COPD).
5. Patients who currently have active pulmonary Tuberculosis
6. Patients who have had eye surgery in the past 3 months or who have a detached retina
7. Patients involved in another interventional asthma study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadians diagnosed with Asthma and 18 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Aaron, MD, Principal Investigator — Ottawa Hosptial Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada